CLINICAL TRIAL: NCT06555848
Title: A Post-Market Prospective Cohort Study on Subjects Receiving CERAMENT G as Part of the Surgical Treatment of Osteomyelitis in a Single-Stage Procedure
Brief Title: CERAMENT G as Part of the Surgical Treatment of Osteomyelitis in a Single-Stage Procedure
Acronym: CERTITUDE
Status: Recruiting | Type: Observational
Sponsor: BONESUPPORT AB (Industry)
Responsible Party: Sponsor
Other Study IDs: 339381
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Osteomyelitis
MeSH Terms: conditions — Osteomyelitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CERAMENT G: Subjects receiving CERAMENT G as part of the surgical treatment of Osteomyelitis
  Interventions: Device: CERAMENT G

INTERVENTIONS:
Device: CERAMENT G — CERAMENT G is intended for use as a bone void filler as an adjunct to systemic antibiotic therapy and surgical debridement (standard treatment approach to a bone infection) as part of the surgical treatment of osteomyelitis. By eluting gentamicin, CERAMENT G can reduce the recurrence of chronic osteomyelitis from gentamicin-sensitive microorganisms in order to protect bone healing.

SUMMARY:
The study is a prospective cohort study of subjects where CERAMENT G was used as part of the surgical treatment of osteomyelitis in a single stage procedure.

DETAILED DESCRIPTION:
The study is a prospective cohort study of subjects where CERAMENT G was used as part of the surgical treatment of osteomyelitis in a single stage procedure.

The purpose of this post market prospective cohort study is to obtain longer-term clinical and radiographic data on the safety and effectiveness of CERAMENT G as part of the surgical treatment of Osteomyelitis in a single-stage procedure.

Detailed questions to be answered are:

1. What is the nature, severity, and frequency of incomplete new bone formation?
2. What is the nature, severity, and frequency of the risks of probable adverse events and serious adverse events associated with incomplete new bone formation, including pathologic fractures and reinfection?

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting the following inclusion criteria are to be included in the analysis:

1. Patients receiving CERAMENT G subsequent to surgical excision of osteomyelitis, with Cierny-Mader classification grades III or IV, who require dead-space management of a bone defect following surgical debridement and excision of infection.
2. Symptoms for a minimum of six months with clinical and radiological features accompanied by at least one of the following:

   1. the presence of a sinus
   2. the presence of an abscess or intra-operative pus
   3. the presence of positive supportive histology
   4. two or more microbiological cultures with indistinguishable organisms (defined as cultures resulting in identification of the same microbe (e.g., Staph aureus) with similar antimicrobial sensitivity) Notes: In cases where cultures are negative, a patient will be included in the study only if there is positive supportive histology combined with the presence of a draining sinus or intra-operative pus. Infected non-unions will be included only if the bone loss is < 1cm after debridement and excision of bone has been performed.

Exclusion Criteria:

The subject will be excluded from the study if:

1. Skeletal immaturity, defined as pre-operative/ screening radiology with evidence of incompletely fused physes. (determined by their previous x-rays which are taken as part of their admission, unrelated to the study)
2. Those unable to give informed consent for inclusion in the trial, or those not willing to be included
3. A known allergy or reaction to gentamicin or calcium sulfate
4. Treatment with a combination of different antibiotic-eluting bone graft substitutes
5. They have a segmental bone defect > 1cm
6. Infection of the spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled post-operatively with Osteomyelitis
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Composite Endpoint | 36 months
  Overall subject success requires all four of the following at 36 months post-op:
  * absence of a reinfection of the original site of osteomyelitis;
  * absence of purulent drainage and wound dehiscence/breakdown
  * absence of a secondary surgical intervention, e.g., grafting or removal of residual CERAMENT G at the original site; and,
  * a lack of serious adverse events associated with incomplete new bone formation, including pathologic fracture of the treated limb
Co-Primary Endpoint | 36 months
  A trend showing increasing new bone formation and decreasing CERAMENT G as determined by a comparison of baseline and interim post-operative timepoint radiographic evaluations out to 36 months post-operative

SECONDARY OUTCOMES:
Radiographic Succcess | 36 months
  Radiographic success at 36 months, defined as CERAMENT G resorption and new bone formation (a minimum of mean void-filling of 74% in the subject population) as determined by comparison of the immediate post-op radiographs to those at 36 months
Clinical Success | 36 months
  Clinical success at 36 months, defined as:
  Maintenance or improvement in function (i.e., no decrease of PRO(s) in the SF-12 score between post-operative and 36 months follow-up)

CONTACTS AND LOCATIONS:
Locations (1):
- Bone Infection Unit, Nuffield Orthopaedic Centtre, Oxford University Hospitals, MHS, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No